CLINICAL TRIAL: NCT05559710
Title: Investigation of the Validity and Reliability of the Kinesthetic and Visual Imagery Questionnaire in Children With Duchenne Muscular Dystrophy
Brief Title: Motor Imagery in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Bora, Physiotherapist, Hacettepe University
Other Study IDs: GO 22/750
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMD Group: Children with Duchenne Muscular Dystrophy (DMD) between the ages of 7 and 18 who have been diagnosed with DMD as a result of genetic testing
- Healthy Controls: Helathy children with similar physical characteristics between the ages of 7 and 8

SUMMARY:
Motor imagery (MI) can be defined as a dynamic process in which the person is mentally stimulated without performing the given motor movement. Studies of imagery; demonstrated that it alters a person's ability to learn, performance skills, and important cognitive skills (self-efficacy, self-confidence, effort, motivation). In recent years, it has been shown that motor imagery techniques are used for therapeutic purposes as a current neurorehabilitation approach and that imagery can have positive effects on improving motor activity and functions. However, it has been reported that the biggest difficulty in the use of imagery techniques is the inability to determine to what extent the individual can perform mental representation of movements. For this reason, it is thought that it is necessary to evaluate the motor imagery ability first in order to identify the patients who are suitable for motor imagery training. The Kinesthetic and Visual Imagery Questionnaire (KVIQ) is a motor imagery questionnaire developed for individuals with limited mobility for different reasons. The questionnaire assesses both the visual and kinesthetic dimensions of motor imagery. of the KVIQ; It has also been shown in the literature that it is a valid and reliable questionnaire that enables the appropriate evaluation of motor imagery in different neurological disease groups such as Multiple Sclerosis, Parkinson's disease, and stroke. However, the literature When examined, no evidence was found about the motor imagery ability of individuals with Duchenne muscular dystrophy (DMD). It is foreseen that KVIQ will be especially suitable for patients with DMD of different functional levels, since all its items have been developed to be applied to people with limited physical mobility or physically disabled people in a sitting position. Therefore, in this study, it is aimed to investigate the validity and reliability of the Kinesthetic and Visual Imagery Questionnaire for patients with DMD.

DETAILED DESCRIPTION:
DMD and age matched healthy individuals will be participate the study between the ages of 7 and 18 years.

Children who cannot cooperate with the physiotherapist adequately and who have had any injury and/or surgery to the lower/upper extremities in the last 6 months will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of DMD confirmed by a genetic test result,
* Be between the ages of 7-18,
* More than 27 (27-35 indicates normal cognitive level) from the Modified Mini Mental Test of children aged 7-15 years to be able to cooperate with the physiotherapist's instructions; Children between the ages of 16-18 get more than 24 points from the Mini Mental State Test (24-30 points indicate no cognitive impairment, 20-23 indicates mild, 10-19 moderate, and below 9 indicates severe cognitive impairment),
* Ability to sit for at least 30 minutes with/without support,
* Volunteering to participate in the study.

Exclusion Criteria:

* Insufficient cooperation with the physiotherapist,
* Any injury and/or surgery to the lower/upper extremities in the last 6 months
* Having any additional neurological/orthopedic problems other than DMD.

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Because DMD is X linked recessive disorder, this disorder is seen in male
Study Population: Duchenne Muscular Dystrophy (DMD), X-linked recessive It is a genetic disease that is inherited and has a prevalence of approximately 1/3600-6000 live male births. The disorder is caused by a mutation in the dystrophin gene located on the X chromosome, resulting in complete or partial absence of the dystrophin protein in the cell membrane, resulting in irreversible progressive loss of functional abilities. The symptoms are manifested by gait disturbance between 3-5 years of age, primarily due to progressive weakness in the proximal muscles. Delayed gait, toe walking, duck-like gait, difficulty climbing stairs and running are early signs of Gower's sign. Gait begins to deteriorate between the ages of 3 and 6, and patients become wheelchair dependent at around 10-12 years of age.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | 15 minutes
  he Kinesthetic and Visual Imagery Questionnaire is a representative tool to assess motor imagery ability. The questionnaire can be used to assess healthy individuals, as well as those with physical disabilities. It allows easy evaluation of motor imagery ability in a sitting position with single joint motions. Furthermore, the questionnaire assesses both visual and kinesthetic dimensions of motor imagery. The questionnaire is not self-administered, rather it is administered by a trained assessor. It assesses the vividness of each dimension of motor imagery (clarity of the image/intensity of sensation) on a 5-point ordinal scale.The long version comprises 20 items (10 movements for each scale) and the short version includes 10 items (5 movements for each scale). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Movement Imagery Questionnaire-Children(MIQ-C) | 20 minutes
  Visual and Kinesthetic motor imagery ability will be evaluated with MIQ-C. Includes 12 items in total. The individual is asked to visualize four different movements from three different imagery perspectives. The clearness of the imagination is scored using a Likert-type scale between 1 (very difficult to feel) -7 (very easy to feel)
Modified Mini Mental Test (MMMT) | 5 minutes
  This test; orientation, memory (recording), attention and calculation, recall and language subtests. The highest score that can be obtained from MMMT is 35. The application time of the test is approximately 5-10 minutes. It has been reported that this test is a suitable tool for the examination of mental functions from the age of 4 and can be easily included in routine neurological examinations of children. Children between the ages of 7 and 15 who get 27 points below the MMMT will be excluded from the study. Children's total score will be recorded
Mini Mental State Test | 5 minutes
  A mini mental state test will be used to evaluate the mental state of children aged 16-18. Test; It evaluates verbal responses including attention, orientation, memory and language skills, ability to obey verbal and written orders, write spontaneous sentences, and copy a complex drawing. The maximum score that can be obtained from the test is 30, the minimum score is 0.
Montreal Cognitive Assessment Scale (MoCA) | 10 minutes
  In this test, which was developed as a rapid screening test for mild cognitive disorders; 8 different cognitive functions are evaluated, including attention, concentration, executive functions, memory, language, visual construction skills, abstract thinking, calculation and orientation. The application time of MoCA, which evaluates abstract thinking in addition to the other test, is approximately 10 minutes. The minimum score that can be taken from the test is 0 and the maximum score is 30. Accordingly, a score of 21 and above indicates normal cognitive functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Bora-Zereyak M, Bulut N, Yilmaz O, Alemdaroglu-Gurbuz I. Motor imagery ability of children with duchenne muscular dystrophy: Reliability and validity of kinesthetic and Visual Imagery Questionnaire-10, and its association with cognitive status. Eur J Paediatr Neurol. 2024 Jul;51:118-124. doi: 10.1016/j.ejpn.2024.06.003. Epub 2024 Jun 15. PMID 38917696